CLINICAL TRIAL: NCT04635371
Title: Monitoring Patients With Acute Cardiac Disease Using a Wireless, Wearable, Non-invasive PPG-based Monitor in the Cardiac ICU
Brief Title: Monitoring Patients With Acute Cardiac Disease Using a Wireless, Wearable, Non-invasive Monitor
Status: Completed | Type: Observational
Sponsor: Biobeat Technologies Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PPGCICUWOMC
Record Dates: First submitted 2020-11-08; First posted 2020-11-19 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Acute Cardiac Event; Acute Cardiac Failure; Acute Cardiac Pulmonary Edema
Keywords: Acute Catdiac Events; Remote Patient Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Non-invasive Monitoring — Wearable, wireless, non-invasive chest-patch devices will be attached to the patients following recruitment and aigning an informed consent form, and from that moment on, vitals will be collected automatically and analyzed retrospectively.

SUMMARY:
A prospective observational study in patients admitted with an acute cardiac disease, in which the PPG-based device will be attached to them on admission, for frequent monitoring of their vitals during hospitalization and interventional procedures. in parallel to currently-used and approved devices. Data will be crossed with gathered clinical and laboratory data, to study the device's ability to detect acute hemodynamic and respiratory changes during hospitalization, and gathering workflow information from the nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and above admitted to the Cardiac ICU due to an acute cardiac event.

Exclusion Criteria:

* Pregnant women, subjects under the age of 18 years.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 men and women admitted to the cardiac ICU with acute caridac event.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Detection of cardio-respiratory changes | Through study completion, an average of 1 year.
  Detection of acute cardio-respiratory/hemodynamic changes during hospitalization and during interventional procedures conducted in the cardiac ICU.

SECONDARY OUTCOMES:
Workflow assessment. | Through study completion, an average of 1 year.
  Nursing staff will be asked - using questionnaires - to assess whether the use of these devices helps in reducing burden of work and increase other interactions with the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Rubinshtein, MD, Principal Investigator — The Edith Wolfson Medical Center
Locations (1):
- The Edith Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: Undecided